CLINICAL TRIAL: NCT02693106
Title: Stimulating the Ketogenesis by Using Nutritional Supplements
Brief Title: Evaluation of the Ketogenic Potential of Different Diet Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-387
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Healthy Adults
Keywords: Ketones; Butyrate; Leucine; Octanoate; Carnitine; Medium Chain Triglycerides
MeSH Terms: conditions — Ketosis | interventions — Leucine; Butyrates; octanoic acid; Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketogenic potential (Experimental): Each participant has to go through a total of 8 visits, each visit corresponding to a standardize breakfast taken alone (control visit) or with one of the dietary supplements evaluated followed by a period of 4-hour with multiple blood sampling.
  Intervention 1: Control; no supplement Intervention 2: 5 g of leucine Intervention 3: 3.6 g of butyrate Intervention 4: 7.2 g of butyrate Intervention 5: 5 g of octanoate Intervention 6: 10 g of octanoate Intervention 7: 1.95 g of carnitine Intervention 8: 65 g of butter fraction rich in MCT
  Interventions: Dietary Supplement: Control; Dietary Supplement: Leucine; Dietary Supplement: Butyrate -; Dietary Supplement: Butyrate +; Dietary Supplement: Octanoate -; Dietary Supplement: Octanoate +; Dietary Supplement: Carnitine; Dietary Supplement: Butter fraction

INTERVENTIONS:
Dietary Supplement: Control — Visit corresponding to a standardize breakfast taken alone (control visit) followed by a period of 4-hour with multiple blood sampling.
  Other Names: CTL
Dietary Supplement: Leucine — Visit corresponding to a standardize breakfast with 5 g of leucine followed by a period of 4-hour with multiple blood sampling.
Dietary Supplement: Butyrate - — Visit corresponding to a standardize breakfast with 3.6 g of butyrate followed by a period of 4-hour with multiple blood sampling.
Dietary Supplement: Butyrate + — Visit corresponding to a standardize breakfast with 7.2 g of butyrate followed by a period of 4-hour with multiple blood sampling.
Dietary Supplement: Octanoate - — Visit corresponding to a standardize breakfast with 5 g of octanoate followed by a period of 4-hour with multiple blood sampling.
Dietary Supplement: Octanoate + — Visit corresponding to a standardize breakfast with 10 g of octanoate followed by a period of 4-hour with multiple blood sampling.
Dietary Supplement: Carnitine — Visit corresponding to a standardize breakfast with 1.95 g of carnitine followed by a period of 4-hour with multiple blood sampling.
Dietary Supplement: Butter fraction — Visit corresponding to a standardize breakfast with 65 g of butter fraction followed by a period of 4-hour with multiple blood sampling.

SUMMARY:
Evaluate the capacity of different dietary supplements to increase ketone production in healthy adults.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the capacity of different dietary supplements to increase ketone production in healthy adults. Each supplement (leucine, butyrate, octanoate, carnitine or butter fraction rich in MCT) is evaluated for a period of 4-hour during which multiple blood samples are taken in order to measure ketone production.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged of 18 years old or older.
* Non-smoking.

Exclusion Criteria:

* Diabetes or prediabetes
* Uncontrolled hypertension
* Uncontrolled thyroid function
* Taking medication that will affect lipid/glucose metabolism
* Severe infection or inflammation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cunnane, PhD, Principal Investigator — Research Centre on Aging CSSS-IUGS - CIUSSS de l'Estrie - CHUS
Locations (1):
- Research Centre on Aging (CSSS-IUGS - CIUSSS de l'Estrie - CHUS), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketogenic Potential
Started | 13
Completed | 10
Not Completed | 3
Not completed — No time | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ketogenic Potential
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 13

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Total Plasma Ketones
Description: Difference from Time 0 in Total ketones = acetoacetate (umol/L) + beta-hydroxybutyrate (umol/L) Time 0 is when the participants arrived, after a 12 hours fast, i.e. before the breakfast.
  Plasma was collected every 30 minutes for 4 hours immediately following breakfast (where supplements were taken).
  Results are the mean of plasma ketones measured every 30 minutes ( i.e. total of 9 plasma samples) for the 4 hour period.
  For each time point, the difference form time 0 has been made. So this is the mean of the difference from time 0 in total ketones.
  Data were not collected for the 'Intervention 8: 65 g of butter fraction rich in MCT' supplement.
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Ketogenic Potential
Number analyzed (Participants) | 10
µmol/L
  CTL | -18.2 (20)
  Leucine | 23 (25)
  Butyrate 3.6g | 12.2 (44.4)
  Butyrate 7.2g | 68.5 (35.9)
  Octanoate 5g | -3.4 (32.8)
  Octanoate 10 g | 39.7 (34)
  Carnitine | -30 (21.4)

ADVERSE EVENTS:
Time Frame: 8 visits of 4 hours
Description: no participants received the intervention if 65 g of butter fraction rich in MCT
Groups:
- Control, no Supplement: Each visit corresponding to a standardize breakfast taken alone (control visit)followed by a period of 4-hour with multiple blood sampling.
- 5g of Leucine: Each visit corresponding to a standardize breakfast taken with 5g of leucine followed by a period of 4-hour with multiple blood sampling.
- 3.6g de Butyrate: Each visit corresponding to a standardize breakfast taken with 3.6g of butyrate followed by a period of 4-hour with multiple blood sampling.
- 7.2g de Butyrate: Each visit corresponding to a standardize breakfast taken with 7.2g of butyrate followed by a period of 4-hour with multiple blood sampling.
- 5g d'Octanoate: Each visit corresponding to a standardize breakfast taken with 5g of octanoate followed by a period of 4-hour with multiple blood sampling.
- 10g d'Octanoate: Each visit corresponding to a standardize breakfast taken with 10g of octanoate followed by a period of 4-hour with multiple blood sampling.
- 1.95g de Carnitine: Each visit corresponding to a standardize breakfast taken with 1.95g of carnitine followed by a period of 4-hour with multiple blood sampling.
Arm/Group | Control, no Supplement | 5g of Leucine | 3.6g de Butyrate | 7.2g de Butyrate | 5g d'Octanoate | 10g d'Octanoate | 1.95g de Carnitine
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 2/10 | 3/10 | 2/10 | 3/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control, no Supplement (N=10) | 5g of Leucine (N=10) | 3.6g de Butyrate (N=10) | 7.2g de Butyrate (N=10) | 5g d'Octanoate (N=10) | 10g d'Octanoate (N=10) | 1.95g de Carnitine (N=10)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
gastric reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Nausea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes